CLINICAL TRIAL: NCT03228823
Title: Prospective Assessment of Premature Ventricular Contractions Suppression in Cardiomyopathy(PAPS): A Pilot Study
Brief Title: Prospective Assessment of Premature Ventricular Contractions Suppression in Cardiomyopathy(PAPS)
Acronym: PAPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); University of California, San Francisco (Other); University of Calgary (Other); Washington University School of Medicine (Other); Wake Forest University Health Sciences (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jose Huizar, Director, Arrhythmia and Device Clinic, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIH ID 9372611; R34HL138110-01 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Ventricular Premature Beats, Contractions, or Systoles; Cardiomyopathies
Keywords: Premature Ventricular contractions; Cardiomyopathy
MeSH Terms: conditions — Ventricular Premature Complexes; Cardiomyopathies | interventions — Radiofrequency Ablation; Amiodarone; Anti-Arrhythmia Agents

STUDY DESIGN:
Intervention Model Description: PVC suppression with either antiarrhythmic drugs or radiofrequency ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Radiofrequency Ablation (Active Comparator): Radiofrequency ablation (RFA) will be performed after 3-month observation period. EPS and RFA will be performed using standard techniques and protocols similar to those patients that do not participate in this clinical study. In the event of polymorphic PVCs, all morphologies are to be targeted for ablation
  Interventions: Procedure: Radiofrequency ablation
- Antiarrhythmic Drug (Active Comparator): Antiarrhythmic drugs (AADs) will be only initiated after 3-month observation period. AAD therapy of choice is amiodarone. Amiodarone loading dose of 10 grams is recommended, followed by maintenance dose of 200-400mg daily to achieve successful PVC suppression. Investigators define successful PVC suppression only if ≥ 80% absolute reduction in PVC burden is achieved after a drug or intervention. Alternatively, sotalol and/or propafenone could be considered at discretion of electrophysiologists (sotalol dose of at least 120mg twice daily, propafenone 150-300mg tid) if there is a significant concern of safety profile of amiodarone.
  Interventions: Drug: Amiodarone (Antiarrhythmic drug)

INTERVENTIONS:
Procedure: Radiofrequency ablation — RFA to achieve PVC suppression will be performed using standard techniques and protocols similar to those patients that do not participate in this clinical study.
  Other Names: Ablation
  Arms: Radiofrequency Ablation
Drug: Amiodarone (Antiarrhythmic drug) — AAD therapy of choice is amiodarone. Amiodarone loading dose of 10 grams is recommended, followed by maintenance dose of 200-400mg daily to achieve successful PVC suppression. Alternatively, sotalol and/or propafenone could be considered at discretion of electrophysiologists (sotalol dose of at least 120mg twice daily, propafenone 150-300mg tid) if there is a significant concern of safety profile of amiodarone.
  Other Names: Amiodarone
  Arms: Antiarrhythmic Drug

SUMMARY:
Premature ventricular contractions (PVCs) coexist in patients with heart failure (HF) and LV dysfunction. Frequent PVCs have shown to induce a reversible cardiomyopathy (PVC-CM).

This clinical pilot study will enroll 36 patients with frequent PVCs (burden >10%) and CM (LVEF <45%) and randomize them to either: 1) RFA or 2) AADs. Prior to treatment, patients will undergo a baseline cardiac MR if clinically indicated followed by 3-month observation period (optimal HF medical therapy). Changes in LV function/scar, PVC burden/arrhythmias and clinical/functional status (QOL, HF symptoms and admissions, NYHA class) and adverse events will be assessed throughout the observation period and compare with PVC suppression strategies (RFA or AAD). Similar comparison will be made between RFA and AAD treatment groups during a 12-month follow up using a Prospective Randomized Open, Blinded End-point (PROBE) study design. The treatment regimens will be compared in an intention-to-treat analysis. In addition, a total of 20,000 consecutive ambulatory ECG Holter monitors from all participating centers will be screened to identify all patients with probable diagnosis of PVC-CM.

This pilot study is intended to estimate the prevalence of this clinical entity and pave the way for a large full scale randomized trial to identify best treatment strategy for patients with PVC-CM. Treating and reversing this underestimated PVC-CM may improve patient's health and subsequently decrease HF healthcare spending.

DETAILED DESCRIPTION:
Rationale. Frequent PVCs have shown to induce a reversible cardiomyopathy (PVC-CM). Yet, it is unclear why some patients develop PVC-CM, while others do not. Appropriate diagnosis and treatment of patients with PVC-CM is believed to carry significant benefits, improving quality of life (QOL), HF symptoms / admissions and life expectancy. Currently, these patients are offered radiofrequency ablation (RFA), antiarrhythmic drugs (AADs) or no treatment depending on physician's experience and resources. Nevertheless, no randomized-prospective study exists to support the benefit of RFA. Thus, a large-scale multicenter randomized clinical trial entitled "Prospective Assessment of PVC Suppression in Cardiomyopathy (PAPS)"' study has been planned to compare these treatment strategies. However, a PAPS pilot study is proposed to better estimate the potential affected patient population, limitations of enrollment, rate of clinical outcomes, potential crossover and drop out. This pilot study is key to better design and power the large-scale multicenter PAPS trial.

Objective. PAPS pilot study is a randomized clinical trial to assess the feasibility of enrolling, randomizing treatment strategies and retaining participants with frequent PVCs and associated CM.

Hypotheses. Our main hypotheses of the PAPS pilot study are:

1. A large-scale randomized PAPS clinical study is feasible with minimal barriers of enrollment, treatment crossover and drop out due to a unique design including a short observation period and PVC suppression strategy in all participants.
2. The rate of responders (defined as improvement of LVEF ≥ 10% points) with HF medical therapy alone during observation period will be less than 15%. In contrast, RFA and AADs will have a responder rate of at least 35% in the same population. Furthermore, RFA will have a greater 1-year response rate when compared to AAD therapy.
3. RFA will have a lower rate of composite adverse events (worsening NYHA class, HF admission, treatment side effects & complications, and death), arrhythmia burden and a better long-term tolerance than AADs.

Methods. A prospective clinical pilot study is planned to prove the feasibility of a large-scale multicenter clinical trial (PAPS study) of patients with probable PVC-CM. This pilot study will enroll 36 patients with frequent PVCs (burden ≥10%) and CM (LVEF ≤45%) and randomize them to either: 1) RFA or 2) AADs. Prior to treatment, all patients will undergo a baseline cardiac MR if clinically indicated and be allowed a 3-month observation period (optimal HF medical therapy). To assess the effects of PVC suppression, changes in LV function, rate of responders (defined above), PVC burden/arrhythmias and clinical/functional status (QOL, HF symptoms and admissions, NYHA class) and adverse events will be compared between observation period and both PVC suppression strategies (RFA or AAD). To identify the best PVC suppression strategy, similar comparisons between RFA and AAD treatment groups will be performed at 12-month follow up using a Prospective Randomized Open, Blinded End-point (PROBE) study design. The treatment regimens will be compared in an intention-to-treat analysis.

In summary, the multicenter PAPS pilot study is intended to better estimate the prevalence of PVC-CM, prove feasibility and rates of clinical outcomes. This pilot study with a multidisciplinary approach will pave the way for a large-scale randomized PAPS trial to identify the best treatment strategy for patients with PVC-CM. Treating and reversing PVC-CM with its associated HF morbidity and mortality will impact not only healthcare spending, but most importantly it will improve patient's health, quality of life and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* LV dysfunction (calculated LVEF < or equal to45% based on Echo) within 150 days of Enrollment (Day 0)
* PVC burden > or equal to 10% by at least a 24-hr ambulatory Holter monitor (within 150 days of Enrollment (Day 0)

Exclusion Criteria:

* Age < 18 years old
* Current amiodarone use or within last 2 months
* Current use of antiarrhythmic drugs class I or III
* Contraindication to amiodarone use or any other class III antiarrhythmic
* Severely symptomatic PVCs (unable to complete 3-month observation period)
* Severe/significant CAD with planned revascularization in the near future
* Complete AV block and pacemaker dependent
* Pacemaker or ICD with >10% RV pacing
* Severe valvular heart disease or planned valvular/cardiac surgery
* Uncontrolled / untreated endocrinopathies
* Uncontrolled HTN, (systolic BP >180mmHg or diastolic >110 mmHg)
* Hypertrophic cardiomyopathy
* Systemic infiltrative and immune disorders
* Family history of dilated CM in a first degree relative
* Alcohol abuse or illicit drug use
* Contraindication to short-term acute anticoagulation (due to possible randomization to ablation)
* Atrial fibrillation and flutter with rapid ventricular response with possible tachycardia-induced cardiomyopathy
* Possible infectious etiology of cardiomyopathy
* Pregnant or lactating women
* Previous PVC ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of left ventricular ejection fraction after PVC suppression | 12 months
  Compare the overall improvement or change in LVEF between RFA and AAD groups.
Responders to PVC suppression strategy | 12 months
  Assessment of the number of responders (delta LVEF ≥ 10%) after PVC suppression strategies will assess the effectiveness of RFA and AADs to reverse or improve cardiomyopathy induced by frequent PVCs.

SECONDARY OUTCOMES:
Successful PVC suppression | 12 months
  Efficacy of Radiofrequency ablation vs. Antiarrhythmic drugs to achieve successful PVC suppression (defined as a reduction of PVC burden greater than ≥80%).
Composite Adverse Events | 12 months
  Composite end-point of adverse events, including worsening in NYHA functional class (I-IV), number of HF and cardiac-related admissions, RFA complications and AAD adverse effects and cardiovascular death.
Composite Arrhythmia Burden | 12 months
  Composite end-point of arrhythmia burden, including PVC recurrence, non-sustained (< 30sec) and sustained (> 30sec) ventricular arrhythmias and arrhythmic sudden cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Jose F Huizar, M.D., Study Director — McGuire VA Medical Center
Locations (11):
- United States (10):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Roxbury VA Medical Center, West Roxbury, Massachusetts
  - Northwell Health System-Staten Island University Hospital, Staten Island, New York
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Libin Cardiovascular Institute, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
This is solely a pilot study of frequent PVCs and cardiomyopathy. Results of this preliminary data will not provide final definitive data, yet investigators will make it available. However, investigators will make clear that this pilot data is not intended to answer benefits of different PVC suppression strategies to avoid misinterpretation or inaccurate conclusions based solely on preliminary data.
Supporting Information: CSR
Time Frame: 3-6 months after pilot study has been completed

REFERENCES:
- [Derived] Torrado J, Sima A, Comstuck C, Kaszala K, Tan A, Koneru J, Frankel DS, Marchlinski F, Kowalski M, Sharma P, Gerstenfeld EP, Vaseghi M, Shivkumar K, Malhotra R, Morillo C, Ellenbogen KA, Huizar JF. Prevalence of frequent premature ventricular contractions and left-ventricular systolic dysfunction in patients receiving Holter monitoring. J Cardiovasc Electrophysiol. 2025 Jan;36(1):54-61. doi: 10.1111/jce.16478. Epub 2024 Oct 24. PMID 39445764

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03228823/Prot_SAP_002.pdf
  • Informed Consent Form (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03228823/ICF_000.pdf